CLINICAL TRIAL: NCT04572958
Title: Changes in Impulse Oscillometry Measurements and Outcomes in Idiopathic Pulmonary Fibrosis
Brief Title: Changes in iOS in IPF
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LO/0969
Record Dates: First submitted 2020-09-26; First posted 2020-10-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a condition where scar tissue (called fibrosis) builds up in the lungs. It usually gets worse over time. Fibrosis causes the lungs to become stiff, and reduces the amount of oxygen that the lungs can take up. People with IPF complain of worsening breathlessness, which limits their day to day activities.

Lung function tests are breathing tests that measure how well your lungs are working, and are used by doctors to decide whether to start or stop medicines in people with IPF. However, people with IPF tell us that lung function tests require a lot of effort, can make them cough and feel very short of breath. About 1 in 5 people with IPF are unable to perform lung function results accurately. This might unfairly lead to some people with IPF not receiving the right medications or for their medications to be stopped too soon.

Impulse oscillometry (iOS) uses sound waves to measure the stiffness of the lung, and has been used successfully in children who are unable to perform normal lung function tests.

The overall aim of the research is to see whether changes in iOS measures can give useful information about the lungs in patients with IPF; for example, by judging the overall impact of the disease on the lungs, or predicting future deterioration.

We will look at how iOS changes over time in patients with IPF, and to see whether these measurements can tell us about whether IPF is getting worse or predict important health events, such as hospital admission. We will compare change in iOS with changes in other tests used to monitor IPF and with patient reported ratings of change in their condition. This will help decide the amount of iOS change that is noticed and considered meaningful by people with IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic pulmonary fibrosis made by specialist multidisciplinary team according to international standards
2. Able to provide written informed consent

Exclusion Criteria:

1. Contraindication to performing conventional lung function tests, e.g untreated TB, haemoptysis, pneumothorax, unstable cardiovascular status, recent eye, thoracic or abdominal surgery, thoracic, abdominal or cerebral aneurysm, acute illness (including diarrhoea and vomiting).
2. Unable to create seal on mouthpiece

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with IPF
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Oscillometry measurements of reactance | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield hospitals, London, Gb-lnd, United Kingdom